CLINICAL TRIAL: NCT04107818
Title: Comparison of Viscoelastic Measurement by ROTEM® Delta and ClotPro® in Trauma Patients. Prospective Observational Study.
Brief Title: Comparison of Viscoelastic Measurement by ROTEM® Delta and ClotPro® in Trauma Patients.
Acronym: ROTCLOT
Status: Completed | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT0022019
Record Dates: First submitted 2019-08-09; First posted 2019-09-27 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Polytrauma; Coagulation Disorder
Keywords: polytrauma; coagulopathy; viscoelastic tests
MeSH Terms: conditions — Multiple Trauma; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to describe the differences and interchangeability in measurements of viscoelastic tests of coagulation by two different devices in adult trauma patients.

DETAILED DESCRIPTION:
The study will commence following the Approval by The Ethics Research Committee. All patients admitted to our emergency department for trauma from the 1st of October 2019 to the 31st of January 2020 will be enrolled after fulfilling the inclusion criteria and in the absence of any exclusion criteria. Informed consent will be requested. Viscoelastic tests of coagulation will be performed on ROTEM® Delta and ClotPro® simultaneously. We will compare values of clotting time (CT), clot formation time (CFT), alfa angle, maximum clot firmness (MCF) and maximum lysis (ML) for test of extrinsic pathway(EX-test) on ClotPro® vs. test for extrinsic pathway (EXTEM) on ROTEM® Delta. Further we will compare values of clotting time (CT), clot formation time (CFT), alfa angle, maximum clot firmness (MCF) and maximum lysis (ML) for thromboelastometry of fibrinogen (FIB-test) on ClotPro® vs. thromboelastometry of fibrinogen (FIBTEM) on ROTEM® Delta. The secondary outcome will be to describe the dependence of measurement on temperature of patient.

Study data will be entered in study form. The measurements can be repeated in time. The indication for next measurement is fully on treating physician.

Differences in estimated viscoelastic coagulation parameters and interchangeability of two devices will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* polytrauma with Injury severity score ≥ 16

Exclusion Criteria:

* pregnancy
* anticoagulant therapy
* antiplatelet therapy
* coagulation disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to emnergency department for severe trauma.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Clotting time (CT) in EX-test and EXTEM | through study completion, an average of 3 months
  difference in clotting time measured by EX-test and EXTEM
Clot formation time (CFT) in EX-test and EXTEM | through study completion, an average of 3 months
  difference in clot formation time measured by EX-test and EXTEM
alfa angle in EX-test and EXTEM | through study completion, an average of 3 months
  difference in alfa angle measured by EX-test and EXTEM
maximum clot firmness (MCF) in EX-test and EXTEM | through study completion, an average of 3 months
  difference in maximum clot firmness measured by EX-test and EXTEM
maximum lysis (ML) in EX-test and EXTEM | through study completion, an average of 3 months
  maximum lysis difference in MCF measured by EX-test and EXTEM
clotting time (CT) FIB-test and FIBTEM | through study completion, an average of 3 months
  difference in clotting time measured by FIB-test and FIBTEM
clot formation time (CFT) FIB-test and FIBTEM | through study completion, an average of 3 months
  difference in clot formation time measured by FIB-test and FIBTEM
maximum clot firmness (MCF) FIB-test and FIBTEM | through study completion, an average of 3 months
  difference in maximum clot firmness measured by FIB-test and FIBTEM
alfa angle FIB-test and FIBTEM | through study completion, an average of 3 months
  difference in alfa angle measured by FIB-test and FIBTEM
maximum lysis (ML) FIB-test and FIBTEM | through study completion, an average of 3 months
  difference in maximum lysis measured by FIB-test and FIBTEM

SECONDARY OUTCOMES:
patient temperature | through study completion, an average of 3 months
  effect of patients´ temperature on results of measurements
maximum clot firmness (MCF) FIB-test and Clauss method | through study completion, an average of 3 months
  correlation of maximum clot firmness with blod fibrinogen level
maximum clot firmness (MCF) FIBTEM and Clauss method | through study completion, an average of 3 months
  correlation of maximum clot firmness with blod fibrinogen level

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, MD., PhD., Study Chair — University Hospital Brno and Masaryk University Brno
Locations (1):
- University Hospital Brno and Masaryk University Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No